CLINICAL TRIAL: NCT07212764
Title: Monitoring Infection Symptoms Through a Mobile Application and Their Effect on Disease Flares in Familial Mediterranean Fever Patients
Brief Title: Mobile App-Based Infection Monitoring in Familial Mediterranean Fever
Status: Enrolling by invitation | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Bengisu Menentoğlu, Principal Investigator, Istanbul University
Other Study IDs: Fmf-Enfeksiyon
Record Dates: First submitted 2025-09-23; First posted 2025-10-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Familial Mediterranean Fever (FMF ); Infection; Mobile Application
Keywords: familial mediterranean fever; mobile application; infection disease
MeSH Terms: conditions — Familial Mediterranean Fever; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FMF group: Patients aged 6-18 years with a diagnosis of FMF according to the Tel Hashomer and Eurofever criteria who agreed to use the mobile application
  Interventions: Other: mobile application

INTERVENTIONS:
Other: mobile application — Patients will be instructed to record any symptoms suggestive of infectious diseases-such as fever, cough, nasal discharge, or myalgia-directly into the mobile application whenever they occur. The app will provide simple checklists and entry fields, allowing patients (or their caregivers) to promptly log these symptoms in real time. By systematically documenting infection-related manifestations alongside routine follow-up data, it will be possible to prospectively evaluate whether infectious episodes act as potential triggers for Familial Mediterranean Fever (FMF) attacks. The collected data will then be analyzed to determine temporal and clinical associations between infection symptoms and subsequent disease flares, thereby clarifying whether infections precipitate or overlap with FMF attacks.

SUMMARY:
Familial Mediterranean Fever (FMF) is an autoinflammatory disease characterized by recurrent episodes of fever, abdominal pain, and serositis. FMF attacks often present with fever and systemic symptoms resembling infectious diseases, making it challenging in clinical practice to distinguish between an attack and an infection. Moreover, infections are known to trigger FMF attacks; however, the number of prospective studies evaluating this association remains limited.

In the current literature, the frequency of attacks and triggering factors in FMF patients have mostly been assessed through retrospective chart reviews. Such methods are prone to incomplete or recall-based data regarding the onset of attacks and infection-related symptoms. With the growing availability of digital health applications, it has become possible to record disease symptoms in real time and on a regular basis, providing more reliable data for both clinicians and researchers.

The present study aims to prospectively evaluate the relationship between infections and disease flares in FMF patients by systematically recording infection symptoms and attack characteristics through a mobile application. This approach is intended to achieve a better understanding of the infection-flare association, improve patient management, and prevent unnecessary treatments. In addition, the feasibility of mobile application-based patient monitoring will be assessed, and its potential contribution to routine clinical practice will be explored.

DETAILED DESCRIPTION:
Infections are well-recognized triggers of FMF attacks; however, the precise relationship between infection episodes and disease flares remains incompletely understood. Most available data on triggering factors have been derived from retrospective chart reviews or patient recall, both of which are prone to incomplete, biased, or delayed reporting. As a result, the temporal dynamics between infection onset and subsequent FMF flares remain insufficiently characterized.

Recent advances in mobile health technologies have created new opportunities to capture disease-related data in real time. Mobile application-based symptom tracking enables patients or caregivers to record clinical events promptly, minimizing recall bias and improving the accuracy and completeness of data collection. This approach facilitates more precise monitoring of the interplay between infections and FMF flares, supports personalized management strategies, and may reduce unnecessary interventions such as unwarranted antibiotic use or hospitalization.

The present study aims to prospectively evaluate the relationship between infections and disease flares in FMF patients using a dedicated mobile application. By systematically recording infection-related symptoms and attack characteristics in real time, the study seeks to: clarify the temporal association between infections and FMF flares; assess the clinical impact of infection-triggered flares on disease course; and evaluate the feasibility and usability of mobile application-based symptom tracking in routine FMF care.

This study is expected to provide more robust evidence on the infection-flare relationship in FMF, refine clinical decision-making during febrile episodes, and contribute to the integration of digital health tools into the routine management of autoinflammatory diseases.

ELIGIBILITY:
Inclusion Criteria

Children and adolescents aged 8-18 years

FMF diagnosis established by Tel Hashomer and/or Eurofever criteria

Regular follow-up at the participating pediatric rheumatology clinic

Stable treatment regimen, defined as:

Colchicine use for ≥ 4 weeks

Biologic or other anti-inflammatory agents stable for ≥ 8 weeks (if applicable)

Access to a smartphone or tablet (iOS/Android) with internet and ability to use the study mobile application (caregiver assistance allowed)

Language proficiency (patient and/or caregiver) sufficient to use the app and respond to prompts

Informed consent from a parent/guardian and assent from the child, as appropriate

Exclusion Criteria

Co-existing chronic inflammatory or autoimmune disorders that may confound flare/infection assessment (e.g., JIA, IBD, Behçet disease) other than FMF

Known primary or secondary immunodeficiency or ongoing immunosuppressive chemotherapy outside standard FMF care

Chronic active infection (e.g., TB, HBV, HCV, HIV) or acute febrile illness at enrollment precluding baseline assessment

Cognitive, visual, or motor limitations preventing app use without caregiver support

No reliable access to a compatible device or internet connection

Concurrent participation in another clinical study likely to affect outcomes or reporting

Anticipated non-adherence (e.g., inability to complete app entries) as judged by the investigator

Refusal or withdrawal of consent/assent

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include children and adolescents aged 6-18 years with a diagnosis of Familial Mediterranean Fever (FMF) according to the Tel Hashomer and/or Eurofever criteria. Participants will be under regular follow-up at the pediatric rheumatology clinic and agree to record infection-related symptoms and FMF complaints through a mobile application. Patients with comorbid chronic inflammatory, autoimmune, or immunodeficiency disorders will be excluded. Informed consent from parents/legal guardians and assent from the child will be obtained.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of FMF Attacks Preceded by Infection-Related Symptoms Recorded via the Mobile Application | 3, 6, 9. months
  Proportion (%) of FMF attacks that occur within 14 days after the onset of infection-related symptoms (fever ≥38 °C, cough, nasal discharge, sore throat, myalgia, etc.) as recorded by patients or caregivers through the mobile application.

SECONDARY OUTCOMES:
Correlation Between Frequency of Infection-Related Symptoms and Frequency of FMF Attacks | 3,6,9. months
  Correlation coefficient (Pearson or Spearman, depending on distribution) between the monthly frequency of infection-related symptoms and the monthly frequency of FMF attacks, based on prospectively recorded data in the mobile application.

CONTACTS AND LOCATIONS:
Overall Officials: Bengisu Menentoğlu, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No